CLINICAL TRIAL: NCT05531643
Title: A Pilot Study of the Safety and Feasibility of Transcutaneous Electrical Nerve Stimulation (TENS) for Chronic Ocular Pain
Brief Title: Pilot Study of TENS for Ocular Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: F3883-P
Record Dates: First submitted 2022-08-30; First posted 2022-09-08 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Eye Pain
Keywords: Eye pain; Dry Eye; Neuropathic Pain; Transcutaneous Electrical Nerve Stimulation
MeSH Terms: conditions — Eye Pain; Dry Eye Syndromes; Neuralgia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants and all study staff involved in participant evaluations will be blinded to treatment allocation. Each device will have the stimulation program pre-set according to the randomization assignment and be numbered. The randomization assignment will be held by the study statistician to match the device number to the intervention assignment. Devices will be distributed in numeric order according to the participant's chronologic order of enrollment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active TENS (Experimental): TENS delivered for 20 minutes to the forehead via the active Cefaly (R) device; at least 3 times per week in-home; for 6 months.
  Interventions: Device: Active Cefaly Dual (R)
- Sham TENS (Sham Comparator): Sham TENS delivered for 20 minutes to the forehead via the sham Cefaly (R) device; at least 3 times per week in-home; for 6 months.
  Interventions: Device: Sham Cefaly Dual (R)

INTERVENTIONS:
Device: Active Cefaly Dual (R) — Transcutaneous electrical nerve stimulation (TENS) device with electrode placement at the forehead. A biphasic rectangular wave will be delivered for a maximum of 20 minutes at a maximum amplitude of 16mA. Participant may halt amplitude before it reaches maximum amplitude. The device has previously been cleared by the FDA for use in migraine patients.
  Arms: Active TENS
Device: Sham Cefaly Dual (R) — Transcutaneous electrical nerve stimulation (TENS) device with electrode placement at the forehead. A 1Hz wave will be delivered for 20 minutes at 1mA.
  Arms: Sham TENS

SUMMARY:
Approximately 20% of Veterans have a diagnosis of dry eye (DE) syndrome which is often accompanied by ocular pain that significantly impacts activities of daily living. Currently very few treatments are available for chronic ocular pain, likely because the mechanisms underlying this type of pain have only recently begun to be studied. New treatments that target the neuropathic mechanisms contributing to this type of pain are needed. The proposed research provides a crucial step in addressing the lack of treatments for neuropathic ocular pain by validating the methodology needed to support a randomized controlled trial of transcutaneous electrical nerve stimulation (TENS). TENS is a non-pharmacologic, non-addictive, non-invasive treatment that has been shown to be effective in other chronic pain conditions. The present pilot study aims to address the need for preliminary support of safety and efficacy of TENS for ocular pain, t to advance the study of new treatments for the long-term relief of chronic ocular pain and its impact on health.

ELIGIBILITY:
Inclusion Criteria:

* male or female
* all races and ethnicities
* at least 18 years of age
* persistent eye pain for at least 6 months
* average eye pain intensity of 4 or more on a 0-10 numerical rating scale
* on a stable medication regimen for at least the past 3 months
* naïve to TENS use for orofacial conditions
* eye pain having neuropathic-like characteristics

Exclusion Criteria:

* presence of ocular diseases that are the likely cause of pain (i.e., corneal and conjunctival scarring, corneal edema, uveitis, iris transillumination defects, etc.)
* contraindication to TENS (i.e., pacemaker, cardioverter defibrillator, neuro-stimulation (brain or spinal cord), bone growth stimulations, indwelling blood pressure monitors, epilepsy, pregnancy)
* patients with confirmed signs of tear dysfunction
* current participation in another study with an investigational drug or device within one month prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Side-effect frequency and severity | 1 year
  An open-ended questionnaire of side-effects will be used to assess any bothersome changes in physical or mental health symptoms every 2 weeks during the 6-month at-home course of treatment. Severity, device/treatment-relatedness of symptoms, and desired or actual discontinuation of device use will be recorded.
Time to peak change in numerical rating scale (NRS, 0-10) | 1 year
  Calculation of time (weeks) to peak reduction in eye pain will be made based on NRS scores obtained every two weeks after initiation of intervention protocol.
Enrollment rate | 1 year
  Percentage of individuals who meet pre-screening requirements, are told about the study, and are consented and enrolled into the study
Screen failure rate | 1 year
  The percentage of individuals who meet pre-screening requirements, consent to study procedures, but who do not meet full criteria after screening visit is conducted
Treatment compliance rate | 1 year
  Calculation of the percentage of individuals who complete at least 75% of treatment session.

SECONDARY OUTCOMES:
Percentage of individuals who score 100% on checklist for proper use of TENS device | 1 year
  The percentage of individuals who, after instruction, score 100% on checklist items for safe and proper use of the device.
Rate of uncertainty in participant treatment allocation guess | 1 year
  Percentage of individuals who rate at least moderate uncertainty in guessing which treatment arm they were allocated to.

OTHER OUTCOMES:
Beta coefficients for participant demographics (sex, age, race/ethnicity) in regression model predicting adherence to treatment protocol | 1 year
  Exploratory regression analysis to identify associations between demographic variables and number of treatment sessions completed
Beta coefficients for participant demographics (sex, age, race/ethnicity) in regression model predicting change in pain (Numerical Rating Scale) | 1 year
  Exploratory regression analysis to identify associations between demographic variables and change in pain ratings (before vs. after 6 month TENS treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth R Felix, PhD, Principal Investigator — Miami VA Healthcare System, Miami, FL
Locations (1):
- Miami VA Healthcare System, Miami, FL, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-02-02): https://cdn.clinicaltrials.gov/large-docs/43/NCT05531643/ICF_000.pdf